CLINICAL TRIAL: NCT04769869
Title: A Single-blind, Randomized, Placebo-controlled 3 Part Study in Healthy Volunteers and Patients With Mild Asthma to Investigate the Safety, Tolerability, and Pharmacokinetics of Inhaled AZD4604 Following Single and Multiple Ascending Doses and to Investigate the Anti-inflammatory Effect of Inhaled AZD4604
Brief Title: A Clinical Trial in Healthy Volunteers and Patients With Mild Asthma to Investigate a New Medicine (AZD4604) for the Treatment of Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: D8210C00001
Record Dates: First submitted 2021-02-12; First posted 2021-02-25 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Asthma
Keywords: AZD4604; Placebo-controlled; Pharmacokinetics; First in Human; Single Ascending Dose; Multiple Ascending Dose; Inhaled Janus Kinase (JAK) Inhibitor
MeSH Terms: conditions — Asthma | interventions — Organization and Administration; Administration, Oral

STUDY DESIGN:
Who Masked: Participant
Masking Description: Part 1a: Healthy volunteers will be blinded to treatment allocation (single-blind design) to minimize bias.
  Part 1b: This part of the study is open-label and blinding is not applicable.
  Part 2: Healthy volunteers will be blinded to treatment allocation (single-blind design) to minimize bias.
  Part 3: Patients will be blinded to treatment allocation (single-blind design) to minimize bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (19):
- Part 1a (SAD): AZD4604 for inhalation via DPI (Dose 1) (Experimental): Healthy volunteers will receive a single inhaled dose of AZD4604 Dose 1 administered with a DPI.
  Interventions: Drug: AZD4604 for inhalation via DPI
- Part 1a (SAD): AZD4604 for inhalation via DPI (Dose 2) (Experimental): Healthy volunteers will receive a single inhaled dose of AZD4604 Dose 2 administered with a DPI.
  Interventions: Drug: AZD4604 for inhalation via DPI
- Part 1a (SAD): AZD4604 for inhalation via DPI(Dose 3) (Experimental): Healthy volunteers will receive a single inhaled dose of AZD4604 Dose 3 administered with a DPI.
  Interventions: Drug: AZD4604 for inhalation via DPI
- Part 1a (SAD): AZD4604 for inhalation via DPI (Dose 4) (Experimental): Healthy volunteers will receive a single inhaled dose of AZD4604 Dose 4 administered with a DPI.
  Interventions: Drug: AZD4604 for inhalation via DPI
- Part 1a (SAD): AZD4604 for inhalation via DPI (Dose 5) (Experimental): Healthy volunteers will receive a single inhaled dose of AZD4604 Dose 5 administered with a DPI.
  Interventions: Drug: AZD4604 for inhalation via DPI
- Part 1a (SAD): AZD4604 for inhalation via DPI (Dose 6) (Experimental): Healthy volunteers will receive a single inhaled dose of AZD4604 Dose 6 administered with a DPI.
  Interventions: Drug: AZD4604 for inhalation via DPI
- Part 1a (SAD): AZD4604 for inhalation via DPI (Dose 7) (Experimental): Healthy volunteers will receive a single inhaled dose of AZD4604 Dose 7 administered with a DPI.
  Interventions: Drug: AZD4604 for inhalation via DPI
- Part 1a (SAD): AZD4604 for inhalation via DPI (Experimental): An additional cohort of healthy volunteers will receive a single inhaled dose of AZD4604 administered with a DPI.
  Interventions: Drug: AZD4604 for inhalation via DPI
- Part 1a (SAD): Placebo for AZD4604 for inhalation via DPI (Placebo Comparator): Healthy volunteers will receive placebo administered with a DPI.
  Interventions: Drug: Placebo for AZD4604 for inhalation via DPI
- Part 1b: AZD4604 for intravenous administration (Experimental): Healthy volunteers will receive a single IV dose of AZD4604 administered as a 20 minute infusion.
  Interventions: Drug: AZD4604 for IV administration
- Part 1b: AZD4604 for oral administration (Experimental): Healthy volunteers will receive a single PO dose of AZD4604.
  Interventions: Drug: AZD4604 for oral administration
- Part 2 (MAD): AZD4604 for inhalation via DPI (Dose 8) (Experimental): Healthy volunteers will receive multiple inhaled dose of AZD4604 administered with a DPI.
  Interventions: Drug: AZD4604 for inhalation via DPI
- Part 2 (MAD): AZD4604 for inhalation via DPI (Dose 9) (Experimental): Healthy volunteers will receive multiple inhaled dose of AZD4604 administered with a DPI.
  Interventions: Drug: AZD4604 for inhalation via DPI
- Part 2 (MAD): AZD4604 for inhalation via DPI (Dose 10) (Experimental): Healthy volunteers will receive multiple inhaled dose of AZD4604 administered with a DPI.
  Interventions: Drug: AZD4604 for inhalation via DPI
- Part 2 (MAD): Placebo for AZD4604 for inhalation via DPI (Placebo Comparator): Healthy volunteers will receive placebo administered with a DPI.
  Interventions: Drug: Placebo for AZD4604 for inhalation via DPI
- Part 3 (MAD): AZD4604 for inhalation via DPI (Dose 9) (Experimental): Patients will receive multiple inhaled dose of AZD4604 administered with a DPI.
  Interventions: Drug: AZD4604 for inhalation via DPI
- Part 3 (MAD): AZD4604 for inhalation via DPI (Dose 10) (Experimental): Patients will receive multiple inhaled dose of AZD4604 administered with a DPI.
  Interventions: Drug: AZD4604 for inhalation via DPI
- Part 3 (MAD): Placebo for AZD4604 for inhalation via DPI (Placebo Comparator): Patients will receive placebo administered with a DPI.
  Interventions: Drug: Placebo for AZD4604 for inhalation via DPI
- Part 3 (PoM): AZD4604 for inhalation via DPI (Dose 9 or Dose 10) (Experimental): Patients will receive multiple inhaled dose of AZD4604 administered with a DPI.
  Interventions: Drug: AZD4604 for inhalation via DPI

INTERVENTIONS:
Drug: AZD4604 for inhalation via DPI — Healthy volunteers will receive AZD4604 administered with a DPI. The dose is expected to be administered between 10 to 45 minutes, depending upon dose. The dose will be administered after an overnight fast of at least 10 hours. Healthy volunteers will be allowed to drink water to prevent dehydration until 1 hour before dosing.
  Arms: Part 1a (SAD): AZD4604 for inhalation via DPI; Part 1a (SAD): AZD4604 for inhalation via DPI (Dose 1); Part 1a (SAD): AZD4604 for inhalation via DPI (Dose 2); Part 1a (SAD): AZD4604 for inhalation via DPI (Dose 4); Part 1a (SAD): AZD4604 for inhalation via DPI (Dose 5); Part 1a (SAD): AZD4604 for inhalation via DPI (Dose 6); Part 1a (SAD): AZD4604 for inhalation via DPI (Dose 7); Part 1a (SAD): AZD4604 for inhalation via DPI(Dose 3); Part 2 (MAD): AZD4604 for inhalation via DPI (Dose 10); Part 2 (MAD): AZD4604 for inhalation via DPI (Dose 8); Part 2 (MAD): AZD4604 for inhalation via DPI (Dose 9)
Drug: Placebo for AZD4604 for inhalation via DPI — Part 1a: An additional cohort of healthy volunteers will receive a placebo administered with a DPI.
  Part 2: Healthy volunteers will receive placebo administered with a DPI. They will receive BID doses on Day 1 to Day 6, and a single dose will be administered on Day 7.
  Part 3: Patients will receive placebo administered with a DPI. They will receive BID doses on Day 1 to Day 9, and a single dose will be administered on Day 10.
  Arms: Part 1a (SAD): Placebo for AZD4604 for inhalation via DPI; Part 2 (MAD): Placebo for AZD4604 for inhalation via DPI; Part 3 (MAD): Placebo for AZD4604 for inhalation via DPI
Drug: AZD4604 for IV administration — Healthy volunteers will receive a single IV dose of AZD4604 administered over 20 minutes. The dose will be administered after an overnight fast of at least 10 hours. Healthy volunteers will be allowed to drink water to prevent dehydration until 1 hour before dosing.
  Arms: Part 1b: AZD4604 for intravenous administration
Drug: AZD4604 for oral administration — Healthy volunteers will receive a single PO dose of AZD4604. The dose will be administered after an overnight fast of at least 10 hours. Healthy volunteers will be allowed to drink water to prevent dehydration until 1 hour before dosing.
  Arms: Part 1b: AZD4604 for oral administration
Drug: AZD4604 for inhalation via DPI — Patients with mild asthma will also receive AZD4604 administered with a DPI. Patients will receive BID doses on Day 1 to Day 9 (morning and evening with 12-hour intervals between doses), and a single morning dose will be administered on Day 10. On Day 1 and Day 10, the morning dose will be administered after an overnight fast of 10 hours. For all other doses, the dose will be administered after a 1-hour fast.
  Arms: Part 3 (MAD): AZD4604 for inhalation via DPI (Dose 10); Part 3 (MAD): AZD4604 for inhalation via DPI (Dose 9); Part 3 (PoM): AZD4604 for inhalation via DPI (Dose 9 or Dose 10)

SUMMARY:
This is a first in human clinical study. Part 1 of the clinical study will assess the safety and tolerability, as well as the single dose pharmacokinetics (PK), of inhaled AZD4604 in healthy volunteers (Part 1a, single ascending dose [SAD]). The single dose administration will be performed with dry powder inhaler (DPI) formulation of AZD4604. When at least 4 cohorts of the SAD part of the study have been completed, AZD4604 will be administered as a single intravenous (IV) or oral (PO) dose to 2 different cohorts of healthy volunteers (Part 1b). The main purpose is to compare the PK between IV, oral and inhaled administration to further characterize the PK properties of AZD4604 by the various administration routes. The results will be used to improve future study design and interpretation. In Part 2 (Multiple ascending dose [MAD]), AZD4604 will be administered at multiple doses (twice daily [BID], 7 days) to healthy volunteers. In Part 3, AZD4604 will be administered at multiple doses to patients with mild asthma at dose levels assessed in Part 2. The multiple-dose administration will be performed with DPI-formulated AZD4604.

DETAILED DESCRIPTION:
Part 1a of the study will be a randomized, single-blind, placebo-controlled, SAD, sequential group design study. Seven inhaled dose levels of AZD4604 are planned to be investigated in cohorts of 8 healthy volunteers, with 6 healthy volunteers randomly assigned to inhaled AZD4604 and 2 healthy volunteers randomly assigned to inhaled placebo in each cohort.

Part 1a will comprise of:

* A Screening Visit within 28 days before dosing.
* A Treatment Period (Day -1 to Day 7, in the Clinical Unit) with a single inhaled dose of AZD4604 or corresponding placebo on Day 1. Although the anticipated systemic exposure and risk for potential adverse systemic effects are considered to be low for AZD4604, healthy volunteers will remain resident at site for additional 6 days of monitoring.
* A Final Assessment on day of discharge.

In Part 1b, AZD4604 will be administered as a single IV or a PO dose to healthy volunteers in order to compare the PK between IV, PO and inhaled administration. Part 1b will be open-label and consist of 2 dose cohorts, IV and PO, with 6 healthy volunteers in each.

Part 1b will comprise of:

* A washout period of at least 2 weeks for the healthy volunteers who received inhaled dosing in Part 1a will occur before IV or PO dosing in Part 1b. All healthy volunteers will have a Screening Visit within 28 days of dosing.
* A Treatment Period (Day -1 to Day 3, in the Clinical Unit) with a single IV or PO dose of AZD4604 on Day 1.
* A Follow-up Visit within 6 ± 1 day after dosing.

Part 2 of the study will be a randomized, single-blind, placebo-controlled, MAD, sequential group design. This part of the study will be conducted in up to 32 healthy volunteers.

Part 2 will comprise of:

* A Screening Visit within 28 days before first dosing.
* A Treatment Period (Day -1 to Day 12 in the Clinical Unit) with twice daily (BID) inhaled doses of AZD4604 or placebo on Day 1 to Day 6 (12-hour [+/- 30 minutes] intervals between doses), and a single inhaled dose on Day 7. The healthy volunteers will remain resident at site for additional 6 days of monitoring, which is predicted to allow sufficient time for near complete washout (estimated time for > 97% of the dose to have been eliminated) of any target engagement from the lungs. Healthy volunteers will remain in the Clinical Unit for the duration of the treatment period and will be discharged on Day 13, 6 days after administration of the last dose.
* A Final Assessment on day of discharge.

Part 3 of the study will be a randomized, single-blind, placebo-controlled, multiple-dose, PK and pharmacodynamic (PD) study part, with daily non-residential visits during the Treatment Period. This part of the study will be conducted in at least 45 patients with mild asthma (16 patients in Cohorts 1 and 2 and at least 29 patients in the Proof of Mechanism [PoM] Cohort).

Part 3 will comprise of:

* A Screening Visit within 42 days before first dosing.
* A Treatment Period (Day -3 to Day 15 as daily non-residential visits) with BID inhaled doses of AZD4604 or placebo on Day 1 to Day 9 (12-hour intervals between doses), and a single inhaled dose on Day 10. Dosing will take place at the clinical site and patients will need to visit the site twice daily on Day 1 to Day 9. The anticipated systemic exposure and risk for potential adverse systemic effects are considered to be low for AZD4604, therefore, patients will not be required to be resident at site during the Treatment Period.
* A Final Assessment (Day 16) on the last day of the Treatment Period.

ELIGIBILITY:
Inclusion criteria:

All Study Parts:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Female subjects must have a negative pregnancy test at the Screening Visit and on admission to the Study Center or prior to randomization for Part 3 (Day -1 or Day 1 visit) and must not be lactating. Women of non-childbearing potential, must fulfill one of the following criteria:

  * Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle stimulating hormone levels in the postmenopausal range.
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not bilateral tubal ligation.
* Male subjects and their Women of childbearing potential (WOCBP) partners should be willing to use highly effective contraception measures and should refrain from donating sperm or fathering a child from the first day of dosing until 3 months after the last dose of investigational medicinal product (IMP).
* WOCBP must be willing to use highly effective contraception measures from the first day of dosing until at least 1 month after the last dose of IMP, such as measures that results in low failure rate, ie, less than 1% per year.

Part 1a, Part 1b, and Part 2 Only:

* Healthy male and female (including WOCBP) volunteers aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture.
* Have a BMI between 18 and 30 kg/m2 inclusive and weigh at least 60 kg.

Part 1a and Part 2 Only:

- Healthy volunteers must have a FEV1 ≥ 80% of the predicted value regarding age, height, gender and ethnicity at the Screening and the Randomization Visits in accordance with American Thoracic Society (ATS)/ European Respiratory Society (ERS) criteria.

Part 3 Only:

* Male and female (including WOCBP) patients with mild asthma aged 18 to 65 years with suitable veins for cannulation or repeated venipuncture.
* Have a BMI between 18 and 35 kg/m2 inclusive and weigh at least 60 kg.
* Physician diagnosed mild asthma for at least 6 months prior to Screening Visit.
* Lung function ≥ 70% predicted for FEV1 at the Screening Visit AND on pre-morning dose Day -1, in accordance with the ATS/ERS criteria.
* Have a FeNO of ≥ 40 ppb at the Screening Visit and at the corresponding clock-time of pre-morning dose on Day-3.
* Must have evidence of up-to-date Coronavirus disease 2019 (COVID-19) vaccination status as per local guidelines.

Exclusion criteria:

All Study Parts:

* History of any clinically important disease or disorder.
* Subject has an increased risk of infection.
* History of cancer within the last 10 years except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated and considered cured.
* Disease history suggesting abnormal immune function.
* Have received any vaccine in the 30 days prior to the first dose.
* Has a body temperature of > 37.7°C on Day-1.
* History or presence of gastrointestinal, hepatic or renal disease.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of Investigational medicinal product (IMP).
* High-sensitivity C-reactive protein > upper limit of normal (ULN) at Screening Visit and on Day -1.
* Any clinically important abnormalities in clinical chemistry, hematology or urinalysis results. Consider appropriate ethnicity adjusted local reference ranges for hematology measurements, when available.
* Abnormal vital signs at the Screening Visit, after 5 minutes supine rest.
* Known or suspected history of drug abuse.
* Current smokers or those who have smoked or used nicotine products.
* History of alcohol abuse or excessive intake of alcohol.
* Positive screen for drugs of abuse or cotinine (nicotine).
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD4604.
* Excessive intake of caffeine containing drinks or food (eg, coffee, tea, chocolate).
* Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of investigational medicinal product.
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study.
* Involvement of any AstraZeneca or study Center employee or their close relatives.
* Subject should not participate in the study if they have any ongoing or recent minor medical complaints that may interfere with the interpretation of study data.
* Subjects who cannot communicate reliably.
* Vulnerable subjects.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12 lead ECG that may interfere with the interpretation of QTc interval changes, including abnormal ST T wave morphology, particularly in the clinical study protocol (CSP) defined primary lead or left ventricular hypertrophy.
* Female subjects who are planning a pregnancy during the study period or within 1 month after the last dose of IMP.

Part 1a, Part 1b, and Part 2 Only:

* Any laboratory values with the deviations at the Screening Visit and on Day 1.
* Persistent or intermittent complete Bundle branch block (BBB), Incomplete bundle branch block (IBBB), or Intraventricular conduction delay (IVCD) with ECG interval measured from the onset of the QRS complex to the J point (QRS) > 110 ms.
* Subjects who have medical dietary restrictions or dietary restrictions which the site are unable to cater for.
* Use of any prescribed or nonprescribed medication during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half life.
* History of any respiratory disorders.
* Clinically significant history of allergic rhinitis/hay fever or anaphylaxis.

Part 3 Only:

* Exacerbation of asthma symptoms and requiring the use of oral or IV steroids, antibiotics, Accident and Emergency visit, or hospital admission.
* Any laboratory values with the deviations at the Screening Visit and on Day -1. Abnormal values may be repeated once at the discretion of the PI: (a)Alanine aminotransferase > 1.25 × upper-limit of normal (ULN); (b)Aspartate aminotransferase > 1.25 × ULN; (c)Total bilirubin > 1.25 × ULN; (d) Creatinine > ULN; (e)Absolute neutrophil count < lower limit of normal (LLN) at the Screening Visit; (f) Absolute lymphocyte count < LLN at the Screening Visit; (g)Hemoglobin < LLN
* Persistent or intermittent complete BBB, IBBB, or IVCD with QRS > 110 ms. Patients with IVCD and QRS <120 ms are acceptable if there is no evidence of eg, ventricular hypertrophy or pre-excitation.
* Use of the following medicines before Screening Visit: Long-acting β2 agonists; Biologics for asthma; Inhaled corticosteroids (ICS) > 500 μg per day of beclometasone dipropionate or equivalent; Any ICS at any dose; Oral or injectable steroids for treatment of asthma or respiratory tract infection; Intranasal steroids; Leukotriene antagonists; Xanthines (excluding caffeine), anticholinergics, or cromoglycate; Short-acting bronchodilator other than for rescue.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Part 1a: Number of healthy volunteers with adverse events (AEs) | From screening (SAEs only) up to Final assessment (Day 7)
  Safety and tolerability of AZD4604 following inhaled administration of single ascending doses to healthy volunteers.
Part 2: Number of healthy volunteers with AEs | From screening (SAEs only) up to Final assessment (Day 13)
  Safety and tolerability of AZD4604 following inhaled administration of multiple ascending doses to healthy volunteers.
Part 1b: Maximum observed plasma (peak) drug concentration (Cmax) | From Day 1 to Day 3
  Cmax of AZD4604 following IV and PO administration of a single dose to healthy volunteers.
Part 1b: Time to reach peak or maximum observed concentration or response following drug administration (tmax) | From Day 1 to Day 3
  tmax of AZD4604 following IV and PO administration of a single dose to healthy volunteers.
Part 1b: Terminal rate constant, estimated by log linear least squares regression of the terminal part of the concentration time curve (λz) | From Day 1 to Day 3
  λz of AZD4604 following IV and PO administration of a single dose to healthy volunteers.
Part 1b: Half life associated with terminal slope (λz) of a semi logarithmic concentration time curve (t1/2λz) | From Day 1 to Day 3
  t1/2λz of AZD4604 following IV and PO administration of a single dose to healthy volunteers.
Part 1b: Partial area under the plasma concentration time curve from time 0 to time 12 (AUC [0 - 12]) | From Day 1 to Day 3
  AUC (0 - 12) of AZD4604 following IV and PO administration of a single dose to healthy volunteers.
Part 1b: Partial area under the plasma concentration time curve from time 0 to time 24 (AUC [0 - 24]) | From Day 1 to Day 3
  AUC (0 - 24) of AZD4604 following IV and PO administration of a single dose to healthy volunteers.
Part 1b: Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) | From Day 1 to Day 3
  AUClast of AZD4604 following IV and PO administration of a single dose to healthy volunteers.
Part 1b: Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | From Day 1 to Day 3
  AUClast of AZD4604 following PO administration of a single dose to healthy volunteers.
Part 1b: Total body clearance of drug from plasma after intravascular administration (CL) | From Day 1 to Day 3
  CL of AZD4604 following IV administration of a single dose to healthy volunteers.
Part 1b: Volume of distribution (apparent) at steady state following extravascular administration (based on terminal phase) (Vz/F) | From Day 1 to Day 3
  Vz/F of AZD4604 following PO administration of a single dose to healthy volunteers.
Part 1b: Volume of distribution following intravascular administration (based on terminal phase) (Vz) | From Day 1 to Day 3
  Vz of AZD4604 following IV administration of a single dose to healthy volunteers.
Part 1b: Dose normalized AUClast, derived by AUClast divided by the dose administered (AUClast/D) | From Day 1 to Day 3
  AUClast/D of AZD4604 following IV and PO administration of a single dose to healthy volunteers.
Part 1b: Area under plasma concentration-time curve from zero to infinity (AUCinf) | From Day 1 to Day 3
  AUCinf of AZD4604 following IV and PO administration of a single dose to healthy volunteers.
Part 1b: Dose normalized AUCinf, derived by AUCinf divided by the dose administered (AUCinf/D) | From Day 1 to Day 3
  AUCinf/D of AZD4604 following IV and PO administration of a single dose to healthy volunteers.
Part 1b: Dose normalized Cmax, derived by Cmax divided by the dose administered (Cmax/D) | From Day 1 to Day 3
  Cmax/D of AZD4604 following IV and PO administration of a single dose to healthy volunteers.
Part 1b: Time of last observed (quantifiable) concentration (tlast) | From Day 1 to Day 3
  tlast of AZD4604 following IV and PO administration of a single dose to healthy volunteers.
Part 3: Number of patients with AEs | From Screening (SAEs only) up to Final Assessment (Day 16)
  Safety and tolerability of AZD4604 following inhaled administration of multiple ascending doses to patients.

SECONDARY OUTCOMES:
Part1b: Number of healthy volunteers with AEs | From screening (only SAEs) to follow-up end of treatment visit (6 ± 1 day post-dose)
  Safety and tolerability of AZD4604 following IV and PO administration of a single dose to healthy volunteers.
Part 1a and Part 2: Cmax | From Day 1 to Day 7 (Part 1a) and from Day 1 to Day 13 (Part 2)
  Cmax of AZD4604 following inhaled administration of single ascending doses and multiple ascending doses of AZD4604 to healthy volunteers.
Part 1a and Part 2: tmax | From Day 1 to Day 7 (Part 1a) and from Day 1 to Day 13 (Part 2)
  tmax of AZD4604 following inhaled administration of single ascending doses and multiple ascending doses of AZD4604 to healthy volunteers.
Part 1a and Part 2: λz | From Day 1 to Day 7 (Part 1a) and on Day 7 (Part 2)
  λz of AZD4604 following inhaled administration of single ascending doses and multiple ascending doses of AZD4604 to healthy volunteers.
Part 1a and Part 2: t1/2λz | From Day 1 to Day 7 (Part 1a) and on Day 7 (Part 2)
  t1/2λz of AZD4604 following inhaled administration of single ascending doses and multiple ascending doses of AZD4604 to healthy volunteers.
Part1a: AUC (0 - 12) | From Day 1 to Day 7
  AUC (0 - 12) of AZD4604 following inhaled administration of single ascending doses of AZD4604 to healthy volunteers.
Part 1a and Part 2: AUC (0 - 24) | From Day 1 to Day 7 (Part 1a) and on Day 7 (Part 2)
  AUC (0 - 24) of AZD4604 following inhaled administration of single ascending doses and multiple ascending doses of AZD4604 to healthy volunteers.
Part 1a and Part 2: AUClast | From Day 1 to Day 7 (Part 1a) and from Day 1 to Day 13 (Part 2)
  AUClast of AZD4604 following inhaled administration of single ascending doses and multiple ascending doses of AZD4604 to healthy volunteers.
Part 2: Area under plasma concentration-time curve in the dose interval (AUCτ) | From Day 1 to Day 13
  AUCτ of AZD4604 following inhaled administration of multiple ascending doses to healthy volunteers.
Part 1a: AUCinf | From Day 1 to Day 7
  AUCinf of AZD4604 following administration of single ascending doses of AZD4604 to healthy volunteers.
Part1a: AUCinf/D | From Day 1 to Day 7
  AUCinf/D of AZD4604 following inhaled administration of single ascending doses of AZD4604 to healthy volunteers.
Part 1a and Part 2: CL/F | From Day 1 to Day 7 (Part 1a) and on Day 7 (Part 2)
  CL/F of AZD4604 following inhaled administration of single and multiple ascending doses of AZD4604 to healthy volunteers.
Part 1a and Part 2: Vz/F | From Day 1 to Day 7 (Part 1a) and on Day 7 (Part 2)
  Vz/F of AZD4604 following inhaled administration of single and multiple ascending doses of AZD4604 to healthy volunteers.
Part 1a and Part 2: AUClast/D | From Day 1 to Day 7 (Part 1a) and from Day 1 to Day 13 (Part 2)
  AUClast/D of AZD4604 following inhaled administration of single and multiple ascending doses of AZD4604 to healthy volunteers.
Part 1a and Part 2: Cmax/D | From Day 1 to Day 7 (Part 1a) and from Day 1 to Day 13 (Part 2)
  Cmax/D of AZD4604 following inhaled administration of single and multiple ascending doses of AZD4604 to healthy volunteers.
Part 1a and Part 2: tlast | From Day 1 to Day 7 (Part 1a) and from Day 1 to Day 13 (Part 2)
  tlast of AZD4604 following inhaled administration of single and multiple ascending doses of AZD4604 to healthy volunteers.
Part 2: Dose normalized AUCτ, derived by AUCτ divided by the dose administered (AUCτ/D) | From Day 1 to Day 13
  AUCτ/D of AZD4604 following inhaled administration of multiple ascending doses to healthy volunteers.
Part 2: Accumulation ratio for AUCτ (Rac AUC) | On Day 7
  Rac AUC of AZD4604 following inhaled administration of multiple ascending doses to healthy volunteers.
Part 2: Accumulation ratio for Cmax (Rac Cmax) | On Day 7
  Rac Cmax of AZD4604 following inhaled administration of multiple ascending doses to healthy volunteers.
Part 1b: Renal clearance of drug from plasma (CLR) | From Day 1 to Day 2
  CLR of AZD4604 following IV administration of a single dose to healthy volunteers.
Part 1b: Cumulative amount of unchanged drug excreted into urine from time t1 to time t2 (Ae [t1 - t2]) | From Day 1 to Day 2
  Ae (t1 - t2) of AZD4604 following IV administration of a single dose to healthy volunteers.
Part 1b: Cumulative percentage of dose excreted unchanged in urine from time t1 to time t2 (fe [t1 - t2]) | From Day 1 to Day 2
  Fe (t1 - t2) of AZD4604 following IV administration of a single dose to healthy volunteers.
Part 2: Cough severity self-assessment (Visual analog scale) | Day-1 to Day 7 (Pre-dose) and Day 8 (Post -dose)
  Effect of AZD4604 on cough severity in healthy will be evaluated volunteers when compared with placebo.
Part 3: Cmax | From Days 1 to 16
  Cmax of AZD4604 following inhaled administration of multiple ascending doses to patients.
Part 3: AUCτ | From Days 1 to 16
  AUCτ of AZD4604 following inhaled administration of multiple ascending doses to patients.
Part 3: AUC | From Days 1 to 16
  AUC of AZD4604 following inhaled administration of multiple ascending doses to patients.
Part 3: Cough severity self-assessment (Visual analog scale) | From Day -3 to -1, and Days 1 to 10
  Effect of AZD4604 on cough severity in patients will be evaluated when compared with placebo.
Part 3: Change from baseline in Fractional exhaled nitric oxide (FeNO) levels | From Day 1 to 10
  Fractional exhaled nitric oxide (FeNO) levels will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Pablo Forte Soto, Principal Investigator — Parexel Early Phase Clinical Unit (London); Rajkumar Chetty, Dr, Principal Investigator — Celerion; Dave Singh, Principal Investigator — Medicines Evaluation Unit; Jorg Taubel, Principal Investigator — Richmond Pharmacology Limited
Locations (3):
- United Kingdom (3):
  - Research Site, Belfast
  - Research Site, Harrow
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please re-refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home